CLINICAL TRIAL: NCT01786915
Title: Phase 1 Randomized, Double-Blind, Placebo-controlled Study of the Safety, Tolerability and Pharmacokinetics of Repeat Administration (7 Days) of Ascending Oral Doses of Bendavia in Healthy Volunteers
Brief Title: Safety and Pharmacokinetic (PK) Study of Oral Bendavia Administered for 7 Days
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: SPIO-102
Record Dates: First submitted 2013-02-06; First posted 2013-02-08 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2014-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — arginyl-2,'6'-dimethyltyrosyl-lysyl-phenylalaninamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bendavia 10mg (Experimental): Bendavia capsule, 10mg, once daily for 7 days
  Interventions: Drug: Bendavia 10mg; Drug: Placebo
- Placebo (Placebo Comparator): Placebo (matching), once daily for 7 days
  Interventions: Drug: Placebo
- Bendavia 50mg (Experimental): Bendavia capsule, 50mg, once daily for 7 days
  Interventions: Drug: Bendavia 50mg; Drug: Placebo

INTERVENTIONS:
Drug: Bendavia 10mg
  Other Names: MTP-131
  Arms: Bendavia 10mg
Drug: Bendavia 50mg
  Other Names: MTP-131
  Arms: Bendavia 50mg
Drug: Placebo

SUMMARY:
The purpose of this study is to assess the study medication blood levels after administration of a repeat oral capsules (one capsule each day for seven days) of Bendavia at one of two dose levels. The effects of Bendavia on the volunteers will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult males or females aged between 18 and 65 years of age with signed informed consent.
* Women who are not post-menopausal (without menstrual bleed for >24 months) or surgically sterile must have a negative serum pregnancy test at screening and within 24 hours of treatment with understanding (through informed consent process) to not become pregnant over the duration of the study and must agree to employ an effective form of birth control for the duration of the study.

  * Acceptable forms of birth control are: double-barrier contraceptives (condom, diaphragm with spermicide) or interuterine device (IUD) 1 week prior to and at least 30 days post treatment even if hormonal contraceptives are used.

Exclusion Criteria:

* Serum sodium level below the lower limit of the site's clinical laboratory normal range at the study qualification visit,
* Clinically significant laboratory abnormalities as determined by the Principal Investigator at laboratory screening
* Creatinine clearance calculated by the Cockcroft and Gault method calculated to be <90 mL/min for males and <80 mL/min for females
* Clinically significant abnormalities on physical examination,
* Body weight less than 60 kg or greater than 80 kg or a body mass index of less than 18 kg/m2 or greater than 32 kg/m2,
* Any disease or condition that might compromise the cardiovascular, hematological, renal, hepatic, pulmonary (including chronic asthma), endocrine (e.g., diabetes), central nervous, or gastrointestinal (including an ulcer) systems,
* History of seizures or history of epilepsy,
* History of serious (Principal Investigator judgment) mental illness,
* Participant in any research involving investigational product within 30 days before planned date of drug administration,
* Positive serology for HIV 1, HIV 2, HBsAg, or hepatitis C virus (HCV),
* Fever greater than 37.5°C at the time of planned dosing,
* Suspicion, or recent history, of alcohol or substance abuse,
* Donated blood or blood products within the past 30 days,
* Women who are pregnant or breastfeeding,
* Employee or family member of an employee of the investigational site,
* Subjects who currently smoke cigarettes, cigars, pipes or chew tobacco products or who have used any tobacco product in the 30 days prior to screening,
* Subjects who are either unwilling to agree to refrain from use or found to be using:

  * Alcohol, caffeine, xanthine-containing food or beverages, nicotine products and over-the-counter medications with the exception of Tylenol from 24 hours prior to dosing and throughout the confinement periods
  * Prescription medications from 14 days prior to and 7 days post treatment (excluding hormonal contraceptives)
  * Hormonal contraceptives without concomitant use of double-barrier contraceptives (condom, diaphragm with spermicide) for a period of 7 days prior to and 30 days post treatment
* Subjects having previous exposure to Bendavia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-02; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Mean peak plasma concentration (Cmax) of Bendavia (ng/ml) on Day 1 in each cohort. | Immediately prior to dosing (Day 1, 0hr) to 24 hours post-dose
  Blood drawn at pre-dose (immediately prior to study drug ingestion) and post-dose at +0.5, +1, +1.5, +2, +2.5, +3, +3.5, +4, +5, +6, +8, +12, +18 hours and pre-Day2-dose (approximately 24 hours post-Day1-dose) will be assessed for Bendavia plasma concentrations. Mean Cmax is defined as the mean of maximum concentration reported for each subject by cohort.
Mean peak plasma concentration (Cmax) of Bendavia (ng/ml) on Day 7 in each cohort. | Immediately prior to dosing (Day 7, 0hr) to 24 hours post-dose
  Blood drawn at Day 7 pre-dose (immediately prior to study drug ingestion) and post-dose at +0.5, +1, +1.5, +2, +2.5, +3, +3.5, +4, +5, +6, +8, +12, +18 and +24 hours will be assessed for Bendavia plasma concentrations. Mean Cmax is defined as the mean of maximum concentration reported for each subject by cohort.
Mean time to peak plasma concentration (Tmax) of Bendavia (hr) on Day 1 in each cohort. | Immediately prior to dosing (Day 1, 0hr) to 24 hours post-dose
  Blood drawn at Day 1 pre-dose (immediately prior to study drug ingestion) and post-dose at +0.5, +1, +1.5, +2, +2.5, +3, +3.5, +4, +5, +6, +8, +12, +18 hours and pre-Day2-dose (approximately 24 hours post-Day1-dose) will be assessed for Bendavia plasma concentrations. Mean Tmax is defined as the mean of the time of maximum concentration reported for each subject by cohort.
Mean time to peak plasma concentration (Tmax) of Bendavia (hr) on Day 7 in each cohort. | Immediately prior to dosing (Day 7, 0hr) to 24 hours post-dose
  Blood drawn at Day 7 pre-dose (immediately prior to study drug ingestion) and post-dose at +0.5, +1, +1.5, +2, +2.5, +3, +3.5, +4, +5, +6, +8, +12, +18 and +24 hours will be assessed for Bendavia plasma concentrations. Mean Tmax is defined as the mean of the time of maximum concentration reported for each subject by cohort.
Mean Area Under the Curve (AUC) from 0-24 hours on Day 1 for Bendavia (hr.ng/ml) in the time from dosing to 24 hours post-dose in each cohort. | Immediately prior to dosing (Day 1, 0hr) to 24 hours post-dose
  Blood drawn at Day 1 pre-dose (immediately prior to study drug ingestion) and post-dose at +0.5, +1, +1.5, +2, +2.5, +3, +3.5, +4, +5, +6, +8, +12 and +18 hours and pre-D2-dose (approximately 24 hours post-D1-dose) will be assessed for Bendavia plasma concentrations. AUC (0-24hr) will be calculated using validated pharmacokinetic analysis software and mean AUC for Bendavia is defined as the mean of AUC (0-24hr) reported for each subject by cohort
Mean Area Under the Curve (AUC) from 0-24 hours on Day 7 for Bendavia (hr.ng/ml) in the time from dosing to 24 hours post-dose in each cohort. | Immediately prior to dosing (Day 1, 0hr) to 24 hours post-dose
  Blood drawn at Day 7 pre-dose (immediately prior to study drug ingestion) and post-dose at +0.5, +1, +1.5, +2, +2.5, +3, +3.5, +4, +5, +6, +8, +12, +18 and +24 hours post-D7-dose will be assessed for Bendavia plasma concentrations. AUC (0-24hr) will be calculated using validated pharmacokinetic analysis software and mean AUC for Bendavia is defined as the mean of AUC (0-24hr) reported for each subject by cohort.
Ratio of AUC0-24h calculated on Day 7 to AUC0-24h calculated on Day 1 [AUC0-24h (d7)/AUC0-24h (d1)]. | Immediately prior to dosing (Day 1, 0hr) to 24 hours post-Day 7-dose
  Mean AUC (0-24hr) calculated at Day 7 as the ratio of Mean AUC (0-24hr) calculated at Day 1 will be calculated for each Bendavia-treated cohort.
Number of adverse events observed with and without Bendavia | From time of study drug administration to End of Study (Day 10)
  Adverse events will be tabulated by treatment group. No statistical analysis will be performed.

SECONDARY OUTCOMES:
Mean change in concentration of urinary 8-isoprostane (pg/mg creatinine) from pre-dose through to study Day 10 for each cohort. | Prior to dosing (Day 1, 0hr) to Study Day 10
  Spot urine samples will be collected at pre-dose on each day of dosing (Days 1-7) and at 24, 48 and 72 hours post-Day7-dose for assay of 8-isoprostane (8-EPIPGF2a) and creatinine. Change from baseline value at each time point assessed will be calculated for each subject. Mean change from baseline is defined as the mean of the change in 8-EPIPGF2a/creatinine for each subject by cohort.
Mean change in concentration of urinary 8-hydroxy-2-deoxyguanosine (ng/mg creatinine) from pre-dose through to study Day 10 for each cohort. | Prior to dosing (Day 1, 0hr) to Study Day 10
  Spot urine samples will be collected at pre-dose on each dosing day (Days 1-7) and at 24, 48 and 72 hours post-D7-dose for assay of 8- hydroxy-2-deoxyguanosine (8-OHDG) and creatinine. Change from baseline value at each time point assessed will be calculated for each subject. Mean change from baseline is defined as the mean of the change in 8-OHDG/creatinine for each subject by cohort.
Mean Area Under the Curve (AUC0-24hr) on Day 1 for Bendavia metabolite M1 (hr.ng/ml) in the time from dosing to 24 hours post-D1-dose in each cohort. | Immediately prior to dosing (Day 1,0hr) to 24 hours post-D1-dose
  Blood drawn at Day 1 pre-dose (immediately prior to study drug ingestion) and post-dose at +0.5, +1, +1.5, +2, +2.5, +3, +3.5, +4, +5, +6, +8, +12, +18 hours and pre-Day2-dose (approximately 24 hours post-Day1-dose) will be assessed for M1 plasma concentrations. AUC (0-24) will be calculated using validated pharmacokinetic analysis software and mean AUC for Bendavia metabolite M1 is defined as the mean of AUC (0-24) reported for each subject by cohort.
Mean Area Under the Curve (AUC0-24hr) on Day 1 for Bendavia metabolite M2 (hr.ng/ml) in the time from dosing to 24 hours post-D1-dose in each cohort. | Immediately prior to dosing (Day 1,0hr) to 24 hours post-D1-dose
  Blood drawn at Day 1 pre-dose (immediately prior to study drug ingestion) and post-dose at +0.5, +1, +1.5, +2, +2.5, +3, +3.5, +4, +5, +6, +8, +12, +18 hours and pre-Day2-dose (approximately 24 hours post-Day1-dose) will be assessed for M2 plasma concentrations. AUC (0-24) will be calculated using validated pharmacokinetic analysis software and mean AUC for Bendavia metabolite M2 is defined as the mean of AUC (0-24) reported for each subject by cohort.
Mean Area Under the Curve on Day 7 (AUC0-24hr) for Bendavia metabolite M1 (hr.ng/ml) in the time from dosing to 24 hours post-D7-dose in each cohort. | Immediately prior to dosing (Day 7,0hr) to 24 hours post-D7-dose
  Blood drawn at Day 7 pre-dose (immediately prior to study drug ingestion) and post-dose at +0.5, +1, +1.5, +2, +2.5, +3, +3.5, +4, +5, +6, +8, +12, +18 and +24 hours will be assessed for M1 plasma concentrations. AUC (0-24) will be calculated using validated pharmacokinetic analysis software and mean AUC for Bendavia metabolite M1 is defined as the mean of AUC (0-24) reported for each subject by cohort.
Mean Area Under the Curve on Day 7 (AUC0-24hr) for Bendavia metabolite M2 (hr.ng/ml) in the time from dosing to 24 hours post-D7-dose in each cohort. | Immediately prior to dosing (Day 7,0hr) to 24 hours post-D7-dose
  Blood drawn at Day 7 pre-dose (immediately prior to study drug ingestion) and post-dose at +0.5, +1, +1.5, +2, +2.5, +3, +3.5, +4, +5, +6, +8, +12, +18 and +24 hours will be assessed for M2 plasma concentrations. AUC (0-24) will be calculated using validated pharmacokinetic analysis software and mean AUC for Bendavia metabolite M2 is defined as the mean of AUC (0-24) reported for each subject by cohort.
Ratio of AUC0-24h for M1 calculated on Day 7 to AUC0-24h calculated on Day 1 [AUC0-24h (d7)/AUC0-24h (d1)]. | Immediately prior to dosing (Day 1, 0hr) to 24 hours post-Day 7-dose
  Mean AUC (0-24hr) for M1 calculated at Day 7 as the ratio of Mean AUC (0-24hr) for M1 calculated at Day 1 will be calculated for each Bendavia-treated cohort.
Ratio of AUC0-24h for M2 calculated on Day 7 to AUC0-24h calculated on Day 1 [AUC0-24h (d7)/AUC0-24h (d1)]. | Immediately prior to dosing (Day 1, 0hr) to 24 hours post-Day 7-dose
  Mean AUC (0-24hr) for M2 calculated at Day 7 as the ratio of Mean AUC (0-24hr) for M2 calculated at Day 1 will be calculated for each Bendavia-treated cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Straube, MD, Study Director — Stealth BioTherapeutics Inc.; Kenneth C Lasseter, MD, Principal Investigator — Climincal Pharmacology of Miami Inc
Locations (1):
- Clinical Pharmacology of Miami Inc, Miami, Florida, United States